CLINICAL TRIAL: NCT03996317
Title: Maternal Hyperoxygenation for Intrapartum Fetal Heart Rate Tracing Abnormalities: a Randomized Clinical Trial
Brief Title: Maternal Hyperoxygenation for Intrapartum Fetal Heart Rate Tracing Abnormalities
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5190191
Record Dates: First submitted 2019-06-18; First posted 2019-06-24 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Perinatal Death; Respiratory Distress Syndrome, Newborn; Hypoxic-Ischemic Encephalopathy; Neonatal Seizure; Meconium Aspiration Syndrome; Intracranial Hemorrhages; Neonatal Hypotension
MeSH Terms: conditions — Perinatal Death; Respiratory Distress Syndrome, Newborn; Hypoxia-Ischemia, Brain; Meconium Aspiration Syndrome; Intracranial Hemorrhages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Standard practice where 10L/min O2 is delivered to patient by mask when any fetal tracing abnormalities are identified.
- Room air (Experimental): O2 will be withheld at times when fetal tracing abnormalities are identified. Patient will continue to breath room air.
  Interventions: Other: Room air

INTERVENTIONS:
Other: Room air — Avoidance of hyperoxygenation
  Arms: Room air

SUMMARY:
Hyperoxygenation for resuscitation of abnormal fetal heart rate tracings has been routine obstetric practice. However, there have not been any studies to support this practice. Recent literature have either found no associated benefit to intrapartum maternal oxygen administration, or in a number of studies demonstrated higher risk of neonatal complications. Despite these studies, the evidences have not been adequate to change the clinical practice because the majority of these studies either focused on biological differences rather than clinical outcomes data or were retrospective rather than randomized trials. Therefore, the investigators propose a large single center randomized clinical trial to determine the effects of maternal hyperoxygenation therapy for the treatment of fetal heart rate tracing abnormalities.

DETAILED DESCRIPTION:
Continuous fetal heart rate tracing is part of the standard practice during intrapartum obstetric management. The goal of fetal heart rate monitoring is to identify early signs of fetal distress during labor, initiate effective interventions to improve fetal outcomes and reduce the risk of cesarean and operative vaginal delivery, and when interventions fail to improve the fetal status, to help guide the decision to proceed with operative delivery in order to minimize fetal/neonatal morbidity as a result of fetal intolerance to labor.

There are four major components to fetal heart tracing that guide obstetric management: baseline, variability, acceleration, and deceleration (uterine contraction pattern is also assessed to guide management). When one or more of these components are outside of normal values, it may be associated with fetal hypoxemia/acidemia. The typical management of these abnormal findings include maternal reposition, IV fluid bolus, increase maternal blood pressure, stopping uterine contractions, amnioinfusion, and maternal oxygen. The goal of therapy is to increase maternal blood flow to the uterus and therefore improve maternal-placental perfusion, increase oxygen delivery to and carbon dioxide removal from the fetus.

Maternal oxygenation is part of the standard management of fetal tracing abnormalities nationwide, and is part of the American College of Obstetricians and Gynecologists (ACOG) guideline for this specific indication. Its use intuitively make sense, as one of the major concerns with fetal tracing abnormalities is the development of fetal hypoxemia leading to anaerobic metabolism and the ensuing development of metabolic acidosis. However, clinical evidence to support its use is lacking. This is partly due to the long-ingrained culture of routine oxygen delivery on Labor and Delivery across the country, therefore no clinical trails were considered until recently. More importantly, from a physiologic standpoint, the fetal hemoglobin has significantly higher oxygen affinity compared to adult hemoglobin. Therefore, increasing maternal oxygen saturation does not lead to significant change in fetal oxygen saturation in general. In addition, some of the reasons for the development of fetal hypoxemia and acidemia are due to placental insufficiency or umbilical cord compression. In these circumstances, there is limited oxygen delivery in the fetal circulation at the maternal-fetal interface and therefore maternal oxygen therapy will have limited effects on fetal oxygenation.

Furthermore, there is growing concern regarding the potential risks associated with supraphysiologic oxygen levels. At a cellular level, hyperoxygenation increased the production of oxygen free radicals, which results in cell damage. This is reflected in the neonatal literature regarding hyperoxygenation during neonatal resuscitation, including higher risk for respiratory and neurologic complications, the American Academy of Pediatrics (AAP) no longer recommend initial neonatal hyperoxygenation during resuscitation. There are similar concerns in oxygen use during obstetric management in recent literature. A number of studies have demonstrated higher risk of neonatal complications associated with maternal intrapartum hyperoxygenation (3-6). However, the evidences have not been adequate to change the clinical practice because the majority of these studies either focused on biological differences rather than clinical outcomes data or were retrospective rather than randomized trials.

Given the ingrained nature of maternal oxygen therapy, the lack of clinical evidence in favor of its use, and concerns regarding potential harm, large scale clinical trials are needed to assess the risks and benefits of the current standard practice. Therefore, the investigators propose a large single center randomized clinical trial to determine the effects of maternal hyperoxygenation therapy for the treatment of fetal heart rate tracing abnormalities.

Trial interventions include the following:

Fetal heart rate abnormalities include one or more of the following:

Recurrent decelerations: more than 2 in a 20 minute period Minimal or absent variability Fetal bradycardia Fetal tachycardia

Routine fetal resuscitation measures will be taken for fetal heart rate abnormalities at the discretion of the obstetric team. These may include:

Maternal repositioning IV fluid bolus Anesthesiology management of hypotension Stopping oxytocin infusion Administering Terbutalin Amnioinfusion Operative vaginal delivery Cesarean delivery In addition to above management options, patient will be assigned to one of two treatment arms through computerized randomization Treatment arm 1 Routine labor management at the discretion of the obstetric team Maternal oxygenation with 10L non-rebreather mask will be given with any above fetal heart rate abnormalities.

Maternal oxygenation is discontinued at the resolution of fetal tracing abnormality or after delivery.

Treatment arm 2 Routine labor management at the discretion of the obstetric team Maternal oxygenation is withheld unless indicated for maternal pulse oximetry is less than 92%

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age between 37and0 weeks and 41and6 weeks
* Admitted for induction of labor or in active labor
* No known fetal anomalies

Exclusion Criteria:

* History of 2 or more cesarean delivery
* Maternal contraindications to labor
* Fetal contraindications to labor
* Maternal hemoglobin <8 on admission
* Maternal medical conditions requiring oxygen supplement at baseline (including but not limited to: severe cardiac conditions, uncontrolled asthma, pulmonary embolism, pulmonary fibrosis, pulmonary edema, pneumonia, sepsis etc.)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal death | Delivery through discharge and average of 1 week
  Death during intrapartum or neonatal period
Respiratory distress syndrome | Delivery through 72 hrs of life
  Need for respiratory support up to 72 hours of life
Low 5 minute Apgar score | At 5 minute of life
  5 minute Apgar score <=3
Hypoxic-ischemic encephalopathy | Delivery through discharge and average of 1 week
Neonatal seizure | Delivery through discharge and average of 1 week
  Seizure or seizure like activity during the neonatal period.
Meconium aspiration syndrome | Delivery through discharge and average of 1 week
Intracranial hemorrhage | Delivery through discharge and average of 1 week
  Intraventricular hemorrhage grades III or IV, subdural hematoma, subarachnoid hematoma, and subgaleal hematoma
Neonatal hypotension | Delivery through discharge and average of 1 week
  hypotension (low average blood pressure) based on weight requiring vasopressor support (medication to increase blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Ruofan Yao, MD MPH, Principal Investigator — Loma Linda University Medical Children's Hospital
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No